CLINICAL TRIAL: NCT00802321
Title: Pharmacokinetic Study of Single Dose Dutasteride in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Jonathan Covault, M.D., Ph.D., University of Connecticut Health Center
Allocation: Randomized | Model: Single Group | Masking: Double
Other Study IDs: 06-217S-2; 620 (Other Grant/Funding Number: GCRC); 5R01AA015606-02 (NIH)
Record Dates: First submitted 2008-12-02; First posted 2008-12-04 (Estimated); Last update posted 2010-09-23 (Estimated); Status verified 2010-09

CONDITIONS: Alcohol Related Disorders; Alcoholism; Alcohol Abuse
Keywords: steroid 5AReductase; genetic polymorphism; GABA receptor
MeSH Terms: conditions — Alcohol-Related Disorders; Alcoholism | interventions — Dutasteride

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (1):
- dutasteride (Experimental)
  Interventions: Drug: Dutasteride

INTERVENTIONS:
Drug: Dutasteride — Subjects will receive a single dose of 2, 3 or 4 mg of dutasteride based on random assignment.
  Other Names: Avodart

SUMMARY:
To monitor the inhibition of 5a-reductase (5AR) enzyme activity at 1, 3, 7, 14, 21, 28 and 42 days following administration of a single dose of dutasteride (2, 3, or 4 mg) by measuring the change in blood levels of 3a-androstanediol glucuronide (3a-diolG) and the ratio of dihydrotestosterone (DHT) to testosterone. To accomplish this aim, an open-label, between-subjects dose comparison study design will be employed with subjects receiving a 2, 3, or 4 mg dosage. Subjects (up to n=40 enrolled to allow a minimum of 24 completers) will be randomly assigned to one of the 3 dose levels. Results of this study will inform the dose selection for a subsequent placebo-controlled, within-subject, crossover study of dutasteride on the effects of alcohol.

A secondary aim of this study is to examine the correlation of a genetic variation in the type I 5AR gene and baseline DHT/T ratio and effect of dutasteride at day 3. A variation in this gene which is one of the targets of dutasteride has been reported to be associated with higher baseline levels of DHT.

DETAILED DESCRIPTION:
Alcohol abuse and dependence remain important public health problems. The chemical mechanisms by which alcohol affects the nervous system are not well understood. Recent theories suggest that alcohol stimulates release of "neuroactive" steroid hormones which are important mediators of alcohol effects. This proposal seeks to identify the most appropriate dosage of an FDA approved medication, dutasteride, which blocks the metabolism of steroid hormones, so that we can use dutasteride as a pharmacologic probe of the biochemistry of alcohol effects in human subjects in a subsequent study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be healthy males volunteers who are 21-55 years old and have a BMI >18.5 and <32.5. All enrolled subjects will have signed IRB approved consent.

Exclusion Criteria:

* Subjects cannot have a current or past DSM-IV diagnosis of alcohol or drug dependence, current or past 12-months diagnosis of alcohol or drug abuse or major psychiatric disorder, neurological illness, have had a hypersensitivity reaction to dutasteride, physical exam evidence of liver dysfunction, currently be using psychotropic medications or medications that are known to influence steroid hormone levels or metabolism. Nicotine-dependent subjects will be excluded to avoid the confounding effects of nicotine withdrawal during day-long laboratory sessions which are part of the planned alcohol administration study as well as effects of tobacco use on metabolism. Subjects who do not agree to use barrier contraception for 1 week after administration of dutasteride will be excluded

Ages: 21 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2006-04; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Change in 5AR enzyme activity as measured by the DHT/testosterone ratio and levels of 3a-androstanediol glucuronide as a function of time after a single loading dose of dutasteride. | 1-42 days

SECONDARY OUTCOMES:
Secondary outcomes include the moderating effect of genetic variation in type I 5AR enzyme on DHT levels and any effects of dutasteride on subjects self report of alcohol use in their everyday life. | 1-42 days

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Covault, M.D, Ph.D, Principal Investigator — UConn Health
Locations (1):
- Unversity of Connecticut Health Center, Farmington, Connecticut, United States